CLINICAL TRIAL: NCT04889781
Title: Piezo-surgery Technique and Intramuscular Dexamethasone Injection to Reduce Postoperative Pain After Impacted Mandibular Third Molar Surgery: A Randomized Clinical Trial
Brief Title: Piezo-surgery Technique and Intramuscular Dexamethasone Injection to Reduce Postoperative Pain After Impacted Mandibular Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Military Healthcare - Oral and Maxillofacial Surgery Department (Other Government)
Responsible Party: Principal Investigator, Wissam Nehme, Head of Oral and Maxillofacial Surgery Department, Central Military Healthcare - Oral and Maxillofacial Surgery Department
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REF 16/02/2019
Record Dates: First submitted 2021-05-09; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Impacted Mandibular Third Molar Extraction
Keywords: Impacted Mandibular Third molar surgery.; Pain; Dexamethasone; Piezosurgery
MeSH Terms: conditions — Pain | interventions — Calcium Dobesilate; Piezosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Rotatory Instruments without Dexamethasone injection (Experimental): Surgical extraction of Impacted Mandibular Third Molar using conventional rotatory instruments to perform osteotomy without Intramuscular Dexamethasone injection
  Interventions: Procedure: Conventional Rotatory instruments
- Rotatory Instruments with Dexamethasone injection (Experimental): Surgical extraction of Impacted Mandibular Third Molar using conventional rotatory instruments to perform osteotomy with 8 mg Intramuscular Dexamethasone injection 30 min before surgery
  Interventions: Drug: Dexamethasone injection
- Piezosurgery technique without Dexamethasone injection (Experimental): Surgical extraction of Impacted Mandibular Third Molar using the piezosurgery technique without Intramuscular Dexamethasone injection
  Interventions: Procedure: Piezosurgery; Procedure: Conventional Rotatory instruments
- Piezosurgery technique with Dexamethasone injection (Experimental): Surgical extraction of Impacted Mandibular Third Molar using the piezosurgery technique with 8 mg Intramuscular Dexamethasone injection 30 min before surgery
  Interventions: Drug: Dexamethasone injection; Procedure: Piezosurgery

INTERVENTIONS:
Drug: Dexamethasone injection — Compare the effect of dexamethasone injection on reducing post-op pain after impacted third molar Surgery
  Arms: Piezosurgery technique with Dexamethasone injection; Rotatory Instruments with Dexamethasone injection
Procedure: Piezosurgery — Compare the effect of Piezosurgery device use on reducing post-op pain after impacted third molar Surgery
  Arms: Piezosurgery technique with Dexamethasone injection; Piezosurgery technique without Dexamethasone injection
Procedure: Conventional Rotatory instruments — Surgical extraction using conventional rotatory instruments to perform osteotomy
  Arms: Piezosurgery technique without Dexamethasone injection; Rotatory Instruments without Dexamethasone injection

SUMMARY:
The purpose of my study is to test the effect of using piezosurgery and dexamethasone injection in the surgical extraction of impacted mandibular third molars, on Postoperative Pain.

DETAILED DESCRIPTION:
Background: Third molar surgery is the most common procedure performed in oral and maxillofacial surgery practice.

This procedure is always associated with varying degrees of postoperative pain and swelling that may have a social impact. Traditionally, rotating instruments like burs have been used for osseous surgery.

Piezosurgery is a novel technique introduced to overcome the disadvantages associated with the conventional rotatory technique. Corticosteroids administration before or after the extraction of third molars is an efficient way to minimize postoperative pain due to their strong anti-inflammatory activity.

Many researchers conducted studies comparing the piezosurgery technique with conventional rotatory technique, regarding postoperative pain and working time, or studies comparing the conventional method with or without dexamethasone injection. Only one recent study (Nov 2018), conducted by Gümrükçü Z. et al. has compared Piezosurgery and dexamethasone injection in third molar surgery, but without evaluating the combined effect of these two techniques on postoperative pain.

Objectives: The objective of this study is to assess the effects of piezosurgery technique and intramuscular dexamethasone injection on postoperative pain in impacted third molar surgery.

Methods: The study design is a randomized controlled clinical trial: 80 patients with mandibular third molar impaction, indicated for surgical extraction should be treated randomly using either the piezosurgery or the conventional rotatory technique, and with or without intramuscular dexamethasone injection. Postoperative pain will be assessed using a visual analog scale (VAS) on days 1, 3, and seven postoperatively.

The differences in Post-operative pain within and between study groups (4 groups) will be tested using repeated measures of analysis of variance (ANOVA) or Friedman tests. Differences in working time among the three techniques will be assessed using a repeated measure of ANOVA. All statistical tests will be two-sided, and the significant level will be set at 0.05. All the analysis will be conducted using the Statistical Package for Social Sciences (SPSS) software version 22.

ELIGIBILITY:
Inclusion Criteria:

* Age from 15 to 30 years,
* Having mandibular impacted third molars,

Exclusion Criteria:

* Heavy smokers (≥20 cigarettes),
* Uncontrolled systemic conditions,
* Infection of the surgery site,
* Psychological problems,
* History of allergy to dexamethasone, amoxicillin, or acetaminophen.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change of Postoperative Pain level From Baseline | Days 1, 3, and 7 Post-op
  Postoperative Pain level using Visual Analogue Scale (VAS): 100 mm in length ranging from 0 for " no pain" to 100 for "the worse imaginable pain
Working time | Per-op
  Surgery time from the start of the incision until the end of the suturing (min).

SECONDARY OUTCOMES:
Change oh The maximal mouth opening From Baseline | At Day 0 and Day 3
  The maximal mouth opening, previously taken at Day 0 was measured at day three post-op, and expressed in millimeters (mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Central Military Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nehme W, Fares Y, Abou-Abbas L. Piezo-surgery technique and intramuscular dexamethasone injection to reduce postoperative pain after impacted mandibular third molar surgery: a randomized clinical trial. BMC Oral Health. 2021 Aug 11;21(1):393. doi: 10.1186/s12903-021-01759-x. PMID 34380473